CLINICAL TRIAL: NCT05830266
Title: Mother-infant Bonding in the Brain: Promoting Maternal Mental Health and High-quality Mother-infant Interactions Via a Mindfulness-based Intervention
Brief Title: Mother-infant Bonding in the Brain: a Mindfulness-based Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tilburg University (Other)
Responsible Party: Principal Investigator, Marion van den Heuvel, Principal Investigator, Tilburg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 222-2022-166
Record Dates: First submitted 2023-03-24; First posted 2023-04-26 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Postpartum Depression; Postpartum Anxiety; Parental Stress
Keywords: Postpartum depression; Postpartum anxiety; Parental stress; Mindfulness; Mindful with your baby; Mother-infant interaction
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "Mindful with your Baby" group-based therapist-guided intervention (Intervention group) (Experimental): Group-based "Mindful with your Baby" therapist-guided intervention via a video-conferencing tool (e.g., Zoom).
  Interventions: Behavioral: "Mindful with your Baby" group-based therapist-guided intervention
- "Mindful with your baby" self-guided online intervention (Waitlist control group) (Other): The waitlist control group receives an individual self-guided online "Mindful with your baby" intervention after a 10-week waiting period.
  Interventions: Behavioral: "Mindful with your baby" self-guided online intervention

INTERVENTIONS:
Behavioral: "Mindful with your Baby" group-based therapist-guided intervention — This 8-sessions long intervention is one of very few interventions that actively includes the baby in the therapy sessions. The intervention includes the following sessions: "Becoming aware of the autopilot", "Practice to really look at your baby", "Getting back in touch with yourself", "Responding sensitively to your baby", "Taking care of yourself in the difficult moments", "Distance and proximity: it's both part of it", "Dealing with expectations of yourself and the environment" and "Mindful parenting: trial and error". The intervention is a group-based therapist-guided intervention via a video-conferencing tool (e.g., Zoom).
  Arms: "Mindful with your Baby" group-based therapist-guided intervention (Intervention group)
Behavioral: "Mindful with your baby" self-guided online intervention — This 8-sessions long intervention includes the following sessions: "Autopilot", "Fresh view", "At home in your body", "Responsive versus reactive parenting", "Kindness to yourself", "Distance and proximity", "Boundaries and taking care of yourself" and "Mindful parenting - day by day". The intervention is an individual self-guided online intervention.
  Arms: "Mindful with your baby" self-guided online intervention (Waitlist control group)

SUMMARY:
The study investigates the effectiveness of the mindfulness-based intervention "Mindful with your Baby" in women with babies between 5-9 months postpartum who experience heightened levels of postpartum depression, anxiety and/or parental stress. The intervention "Mindful with your Baby" is one of the very few interventions for maternal postnatal mental health issues that takes the bond between mother and infant into account. It is hypothesized that the "Mindful with your Baby" intervention will reduce levels of postpartum depression, anxiety and parental stress, and improve mother-infant behavioral interaction and increase neural synchrony between mother and infant brains.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (18+y).
* First antenatal visit < 12 weeks.
* Score above cut off on the Edinburgh Postnatal Depression Scale (EPDS), the anxiety subscale of the Symptom Checklist (SCL-90) and/or the Parental Stress Questionnaire (PSQ) at 8-10 weeks postpartum.
* Dutch-speaking or understanding Dutch.

Exclusion Criteria:

* Gemelli pregnancy (or higher order pregnancy).
* Known endocrine disorder before pregnancy (diabetes-I, Rheumatoid arthritis).
* Severe psychiatric disease (schizophrenia, borderline or bipolar disorder).
* HIV.
* Drug or alcohol addiction problems.
* Any other disease resulting in treatment with drugs that are potentially adverse for the fetus and need careful follow-up during pregnancy.
* No access to the internet.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline postpartum depressive symptoms | before the intervention (baseline, week 0), halfway through the intervention (week 4), post-intervention (week 8) and after 10-weeks follow-up (week 18)
  Assessed with the 10-item Edinburgh Postnatal Depression Scale (EPDS). The EPDS is the most widely used self-rating scale to assess depressive symptoms in the perinatal period. The EPDS total score ranges from 0 to 30, with higher scores indicating more depressive symptoms. The questionnaire has been validated in Dutch postpartum women.
Change from baseline postpartum anxiety symptoms | before the intervention (baseline, week 0), halfway through the intervention (week 4), post-intervention (week 8) and after 10-weeks follow-up (week 18)
  Assessed with the 10-item anxiety subscale of the Symptom Checklist (SCL-90). The total scores range from 10 to 50 and higher scores reflect more anxiety symptoms. The questionnaire has showed good reliability and validity in non-pregnant samples.
Change from baseline parental stress | before the intervention (baseline, week 0), halfway through the intervention (week 4), post-intervention (week 8) and after 10-weeks follow-up (week 18)
  Assessed with the Parental Stress Questionnaire (PSQ, in Dutch: Opvoedingsbelastingvragenlijst), which is based on the Parenting Stress Index. This study uses only the first three subscales related to parenting: parent-child relationship problems, parenting problems and parental role restriction. Total scores range from 19 to 76 with higher scores indicating more parental stress. In order to interpret the level of parental stress experienced, subscale scores are converted into T-scores conform the norms of the child's age (e.g., 0 to 3 years). The questionnaire and subscales have showed good reliability and validity.
Change from baseline mother-infant bonding | Before the intervention (baseline, week 0) and post-intervention (week 8)
  Assessed with video coding
Change from baseline neural synchrony between mother and infant (EEG outcome 1) | Before the intervention (baseline, week 0) and post-intervention (week 8)
  Assessed with dual-EEG, with the Phase Locking Value (PLV) in the alpha band frequency (6-9 Hz) during the free play task. We expect that neural synchrony between mother and infant will increase (more) in the intervention group.
Change from baseline neural synchrony between mother and infant (EEG outcome 2) | Before the intervention (baseline, week 0) and post-intervention (week 8)
  Assessed with dual-EEG, with the Phase Locking Value (PLV) in the alpha band frequency (6-9 Hz) during the still face paradigm. We expect that neural synchrony between mother and infant will increase (more) in the intervention group.

SECONDARY OUTCOMES:
Change from baseline postpartum-specific anxiety | before the intervention (baseline, week 0), halfway through the intervention (week 4), post-intervention (week 8) and after 10-weeks follow-up (week 18)
  Assessed with the 12-item Postpartum Specific Anxiety Scale - Research Short Form - for global Crises (PSAS-RSF-C). Total scores range from 0 to 36, with higher scores representing greater postpartum-specific anxiety. The PSAS-RSF-C has been validated in postpartum women.
Change from baseline worry | before the intervention (baseline, week 0), halfway through the intervention (week 4), post-intervention (week 8) and after 10-weeks follow-up (week 18)
  Assessed with the 16-item Penn-State Worry Questionnaire (PSWQ). The total score ranges from 16 to 80, with higher scores reflecting a stronger tendency to worry. The PSWQ has been validated in Dutch samples.
Change from baseline mindfulness skills | before the intervention (baseline, week 0), halfway through the intervention (week 4), post-intervention (week 8) and after 10-weeks follow-up (week 18)
  Assessed with the 15-item Three Facet Mindfulness Questionnaire Short Form (TFMQ-SF), consisting of the facets acting with awareness, non-judging and non-reacting. The total score ranges from 0 to 60, with higher scores indicating better mindfulness skills. The validity of the measure is established and indices of internal reliability were found to be adequate.
Change from baseline self-compassion | before the intervention (baseline, week 0), halfway through the intervention (week 4), post-intervention (week 8) and after 10-weeks follow-up (week 18)
  Assessed with the 3-item Self-Compassion Scale (SCS-3), which was derived from the Self-Compassion Scale (SCS) and the Self-Compassion Scale Short Form (SCS-SF). The total scores range from 3 to 15, with higher scores indicating higher levels of self-compassion.
Change from baseline bonding | before the intervention (baseline, week 0), halfway through the intervention (week 4), post-intervention (week 8) and after 10-weeks follow-up (week 18)
  Assessed with the 5-item Pre- and Postnatal Bonding Scale (PPBS). Total scores range from 14 to 56, with higher scores reflecting more positive feelings of bonding. The scale has shown good psychometric properties in Dutch perinatal women.
Change from baseline infant temperament | Before the intervention (baseline, week 0), post-intervention (week 8) and after 10-weeks follow-up (week 18)
  Assessed with the Infant Behavior Questionnaire - Revised - very short form (IBQ-R-vsf), including the subscales surgency, negative affect and effortful control. Total scores can be calculated over the items that received a numerical response, and range from 0 to 259. Higher scores reflect greater levels of infant temperament. The IBQ-R-vsf has been validated in parent samples.
Change from baseline mindful parenting | before the intervention (baseline, week 0), halfway through the intervention (week 4), post-intervention (week 8) and after 10-weeks follow-up (week 18)
  Assessed with the 27-item adapted Interpersonal Mindfulness in Parenting Scale (IM-P). Total scores range from 27 to 135, with higher scores indicating greater levels of mindful parenting.
Change from baseline parenting self-efficacy | before the intervention (baseline, week 0), halfway through the intervention (week 4), post-intervention (week 8) and after 10-weeks follow-up (week 18)
  Assessed with the 16-item Maternal Self-Efficacy in the Nurturing Role questionnaire (SENR), of which validity and reliability has been established. Total scores range from 16 to 112, with higher scores representing higher levels of parenting self-efficacy.
Change from baseline personal goal | before the intervention (baseline, week 0), halfway through the intervention (week 4), post-intervention (week 8) and after 10-weeks follow-up (week 18)
  Assessed with Goal Attainment Scaling (GAS). Before the intervention, mothers are asked to write down an overall goal. They also formulate the situation if things are: worse than at the current moment (-1), according to the current moment (0), a little better than the current moment (+1), much better than the current moment (+2), the best possible outcome (+3). In the next assessments, women will see their previously established goal and scales (-1, 0, +1, +2 and +3). They are asked to indicate what describes their current situation best. Validity and reliability of the GAS have been established.

CONTACTS AND LOCATIONS:
Overall Officials: Marion I van den Heuvel, PhD, Principal Investigator — Tilburg University
Locations (1):
- Tilburg University, Tilburg, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No